CLINICAL TRIAL: NCT06156462
Title: A Study Evaluating the Use of ResAppDx v2.0 as an Aid to Diagnose Respiratory Disease in Adolescent and Adult Patients in an Emergency Department
Status: Completed | Type: Observational
Sponsor: ResApp Health Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: 19003
Record Dates: First submitted 2023-11-26; First posted 2023-12-05 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Asthma Exacerbation; COPD Exacerbation; Lower Respiratory Disease; Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Adults: >18 yo
  Interventions: Device: ResAppDx v.20
- Adolescents: <16 yo
  Interventions: Device: ResAppDx v.20

INTERVENTIONS:
Device: ResAppDx v.20 — Software device measuring cough sounds to aid diagnosis of respiratory diseases

SUMMARY:
Aim is to to demonstrate that the ResAppDx v2.0 algorithms provide an accurate diagnosis of respiratory disease in the study's clinical setting compared to a clinical adjudication committee's (CAC) diagnosis; and to establish a baseline for the resource use and cost of current care pathways for respiratory disease diagnosis in an emergency department. Eligible subjects will be consented/enrolled and their subject reported signs/symptoms of respiratory disease will be recorded in the study electronic case report form (eCRF). The enrolled subject's cough sounds will be captured (5 cough sounds are required) using the ResAppDx v2.0 Investigational Device (ID) software installed on a study smartphone; cough sounds may be voluntary and/or involuntary/spontaneous. As this is an observational study the treating team will be blinded to the ResAppDx v2.0 diagnoses. Additional medical information will be collected from the treating team, from the subject and from the subject's medical record. No follow-up/subsequent visits with the subject will be required by the study. As an efficacy comparator, a clinical adjudication committee (CAC) will determine the final clinical diagnosis using the disease case definitions, eCRF data and the subject's medical record. Information on time and scope of tests and consults ordered by the treating team will be recorded to set a baseline for resource use and cost of current standard of care treatment/assessment procedures. This data will allow future health economics analyses to be performed. The blinded ResAppDx v2.0 diagnoses will be unblinded after database lock and sensitivity and specificity will be calculated for the ResAppDx v2.0 diagnoses compared to agreement with the CAC's final clinical diagnoses.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents and adults aged 12 years and older:

  1. Presenting to the study site with current signs or symptoms of rhinorrhea, cough, wheeze, stridor, increased work of breathing, cyanosis, additional auscultatory noises (crepitations), or low oximetry levels.
  2. Onset of symptoms must have occurred within 14 days of presenting to the site.

Exclusion Criteria:

* 1. Parent or legal guardian is unwilling or unable to sign the study informed consent form.

  2. Adolescent patient who, in the opinion of the investigator, is able to provide assent based on their age, maturity or psychological state is unwilling or unable to sign the study assent form.

  3. Patient requires mechanical ventilatory support (including invasive, CPAP, or BiPAP) or high flow nasal cannula.

  4. Patient has a history of structural airways abnormalities, tracheobronchomalacia, or vocal cord abnormalities (e.g. laryngomalacia, tracheomalacia, or bronchomalacia).

  5. Patient has any medical contraindication to voluntary cough, including the following (only enroll if coughing spontaneously):

  a. Severe respiratory distress b. History of pneumothorax c. Eye, chest, or abdominal surgery within 3 months of presenting to the site 6. Hemoptysis within 1 month of presenting to the site. 7. Patient is too medically unstable to participate in study at the discretion of the treating clinician.

  8. Patient has a tracheostomy present and/or has a tracheostomy tube placed. 9. Patient is unable to provide at least 5 coughs (voluntary and/or spontaneous).

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Subjects aged 12 years and older presenting to a study site with signs or symptoms of respiratory disease including rhinorrhea, cough, wheeze, stridor, increased work of breathing, cyanosis, additional auscultatory noises (crepitations), or low oximetry levels.
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Efficacy of ResAppDx v2.0 when compared to clinical adjudication panel | 6 months
  Efficacy will be compared to the diagnosis formed by consensus of the clinical adjudication committee and evaluated using sensitivity and specificity of ResAppDx v2.0 algorithms ("Index Test") to diagnose and rule out the following conditions:
  * Asthma exacerbation;
  * COPD exacerbation;
  * Lower respiratory tract disease (LRTD); and
  * Pneumonia (including lower respiratory tract infection).

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Addenbrookes Hospital, London
  - The Royal London Hospital, London
  - University College London Hospital, London

IPD SHARING:
Plan to Share IPD: No
No IPD available to other researchers